CLINICAL TRIAL: NCT06256731
Title: ETNA-MS Device Validation Study
Acronym: ETNA-MS
Status: Recruiting | Type: Observational
Sponsor: Innodem Neurosciences (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Other Study IDs: IN-MS-001
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort of MS patients with EDSS 1.0-4.5: Confirmed diagnosis of MS with an EDSS score ranging from 1.0 and 4.5.
  Interventions: Device: Eye-Tracking

INTERVENTIONS:
Device: Eye-Tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
The overarching goal of this research protocol is to validate the effectiveness of Innodem's ETNA-MS device in informing clinicians on the disability status of Multiple Sclerosis (MS) patients. Effectiveness of the device will be assessed by the level of agreement between the EDSS estimated by the device and the actual scores measured by the neurologist in-person assessments.

DETAILED DESCRIPTION:
This study will use a multi-site cross-sectional design in a single cohort of Multiple Sclerosis (MS) patients. Eligible patients with MS will be selected and categorized based on their Expanded Disability Status Scale (EDSS) score. Patients eye movements will be captured using the patented eye-tracking technology at one single time point. In addition to the eye-tracking tests, patient phenotypes will be further detailed via brief functional and cognitive assessments using the EDSS, Brief International Cognitive Assessment for MS (BICAMS) and Multiple Sclerosis Functional Composite (MSFC). All patients will be required to participate in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Aged 18 years or older at the time of enrolment
* Able to read in either English, Spanish or French
* Able to read the oculomotor task on-screen instructions at the testing distance (45 cm) with or without corrective lenses
* Confirmed diagnosis of MS as per the Macdonald criteria, irrespective of MS subtype (relapsing-remitting (RRMS), secondary-progressive (SPMS), primary-progressive (PPMS), and progressive-relapsing (PRMS))
* Neurologist-determined EDSS score between 1.0-4.5

Exclusion Criteria:

* Evidence or medical history of a neuropsychiatric disorder such as schizophrenia and autism, which are known to impair eye movements and oculomotor control.
* Presence of comorbid neurological conditions causing significant eye movement anomalies (such as strabismus, cranial nerve palsy, stroke-causing hemianopsia).
* Diagnosis of macular edema or other pre-existing ocular conditions that would prevent a participant from performing the eye movement assessments.
* Having started a new prescription medication or having changed the dose of a medication known to influence ocular motor visual function (e.g. benzodiazepines, antipsychotics, and anticonvulsants) within the past three months.
* Participants with non-disease related physical impairments to a leg, hand, or arm (e.g., broken bone or severe sprain) that would not allow completion of the assessments.
* Having an EDSS score for which the desired sample size has been reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target sample size for the MS group is 60. Eligible patients with MS will be selected and categorized based on their EDSS score.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Validate the effectiveness of the ETNA-MS device to estimate MS disease severity/status as estimated by the EDSS. | Day 1
  Evaluate the average level of agreement (within +/- 0.5 EDSS score) between the device-estimated EDSS score and the ground truth, that is the true EDSS score as established by a certified neurologist. The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.

SECONDARY OUTCOMES:
Validate that the ETNA-MS device has good test-retest reliability for estimating the EDSS. | Day 1
  Evaluate the level of agreement between device outputs from two repeated eye-tracking tests.
Validate the effectiveness of the ETNA-MS device to estimate the Symbol Digit Modalities Test (SDMT) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  Evaluate the level of agreement between the device-estimated clinical scores and the ground truth scores, and between the device-estimated composite scores and the ground truth composite scores. The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the Symbol Digit Modalities Test (SDMT). The test presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Patients are asked to voice or write the digit associated with each symbol as rapidly as possible for 90 seconds. The test is scored on the number correct answers over the 90 second time span. A higher score represents lower levels of disability.
Validate the effectiveness of the ETNA-MS device to estimate the Brief Visuospatial Memory Test-Revised (BVMT-R) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  Evaluate the level of agreement between the device-estimated clinical scores and the ground truth scores, and between the device-estimated composite scores and the ground truth composite scores. The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the Brief Visuospatial Memory Test-Revised (BVMT-R). In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. Thus, scores range from 0 to 12. There are three learning trials, and the test is scored on the total number of points earned over the three learning trials. A higher score represents lower levels of disability.
Validate the effectiveness of the ETNA-MS device to estimate the Rey Auditory Verbal Learning Test (RAVLT) as part of the Brief International Cognitive Assessment for MS (BICAMS). | Day 1
  Evaluate the level of agreement between the device-estimated clinical scores and the ground truth scores, and between the device-estimated composite scores and the ground truth composite scores. The Brief International Cognitive Assessment for MS (BICAMS) is a battery of tests recommended by multiple sclerosis (MS) experts to monitor MS-related cognitive impairment, which includes the Rey Auditory Verbal Learning Test (RAVLT). In this test, patients listen to a 15-word list and report as many of the times as possible. There is no instruction as to the order in which items are recalled. After recall is recorded, the entire list is read again followed by a second attempt at recall. Altogether, there are five learning trials. The test is scored on the total number of recalled items over the five learning trials. The delayed recall, second list, and recognition trials are not administered in the context of this study. A higher score represents lower levels of disability.
Validate the effectiveness of the ETNA-MS device to estimate the Timed 25-foot walk as part of the Multiple sclerosis functional composite (MSFC). | Day 1
  Evaluate the level of agreement between the device-estimated clinical scores and the ground truth scores, and between the device-estimated composite scores and the ground truth composite scores. The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. The test is scored on the time taken to walk the two trials of the 25 feet walk. A higher score represents higher levels of disability.
Validate the effectiveness of the ETNA-MS device to estimate the 9-Hole Peg Test (9-HPT) as part of the Multiple sclerosis functional composite (MSFC). | Day 1
  Evaluate the level of agreement between the device-estimated clinical scores and the ground truth scores, and between the device-estimated composite scores and the ground truth composite scores. The 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice (two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand). The test is scored on the time taken to complete each trial for each hand. A higher score represents higher levels of disability.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - MS Integrated Center, Phoenix, Arizona
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Premier Neurology Research, P.C., Greenville, South Carolina
  - Rocky Mountain MS Research Group, Salt Lake City, Utah